CLINICAL TRIAL: NCT01660685
Title: Effects of Journaling on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Chief, Division of General Internal Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39952EP
Record Dates: First submitted 2012-08-01; First posted 2012-08-09 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Overweight; Obese
Keywords: Weight loss; Web-based; Journaling; Body Mass Index between 27 and 45
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tracking + Journaling + Website (Experimental): In addition to standard care, participants will complete daily tracking and journaling and receive weekly feedback based on their individual entries.
  Interventions: Behavioral: Tracking; Behavioral: Journaling; Behavioral: Website; Behavioral: Enhanced Usual Care
- Enhanced Usual Care (Active Comparator): Participants receive standard care
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Tracking — Participants will record their daily weight, physical activity steps and meal replacements online
  Arms: Tracking + Journaling + Website
Behavioral: Journaling — Participants will journal to two online writing prompts: one on positive focus and one on goal setting
  Arms: Tracking + Journaling + Website
Behavioral: Website — Participants will have access to resource website with stories and tips from people who successfully lost weight, blogs from investigators, quotes from other participants.
  Arms: Tracking + Journaling + Website
Behavioral: Enhanced Usual Care — Participants will receive standard care of monthly height, weight and blood pressure measurements. Participants will also receive a pedometer and a diet plan book on pre-portioned items.

SUMMARY:
This is a randomized controlled trial with enhanced usual care treatment control. The aim is to determine the effects of journaling and use of resource website on weight loss. There will be two groups of 55 participants each. The intervention condition will be asked to record daily weight, physical activity steps taken and pre-portioned food items and to complete two daily journaling activities. Participants will also receive weekly tracing data, a weekly blog from the principal investigator and have access to a weight control website. The control group will not have access to the tracking, journaling or website for three months. Investigators hypothesize that a website paired with tracking and journaling will be more effective in helping participants lose weight.

DETAILED DESCRIPTION:
Participants will call study line given on recruitment materials and be screened over the phone.

Baseline visit:

Individuals who meet the screening criteria will be invited to a one-hour training session about the website and diet plan book. During the training, a coordinator will review the consent form with the participants and ask if they have any questions. The coordinator will take consented individuals' height, weight and blood pressure measurements. Participants will be given a pedometer to use during physical activities and a meal replacement book to use as a resource.

After baseline visit:

All participants will complete surveys online (Demographics, Three-Factor Eating Questionnaire, Motivation, Weight Loss Habits, Medication log, International Physical Activity Questionnaire) and be randomized into one of two groups. The intervention group will be asked to record their weight, physical activity steps, pre-portioned food items and journal entries on a daily basis. The control group will be sent an email informing them they will have access to the tracking, journals and website in three months.

Intervention Group:

Participants will receive daily emails with links to record their weight, physical activity steps and pre-portioned food items; participants will also complete a journaling response to two writing prompts. The emails will contain links to the website to be used as a resource. Every week, participants will enter whether they have an appointment with primary care provider in the next week. Participants will also receive weekly blogs from the principal investigator; participants can opt out of receiving the blog emails at any time. Coordinators will review the database weekly. If a participant has lost ten pounds, they will be emailed to call their doctor since weight loss can affect blood pressure and medication needs. If a participant has an upcoming primary care provider appointment, they will be emailed to print out their tracking graphs (weight, steps taken, meal replacements). Coordinators will also monitor journal responses; coordinators will contact participants who wrote useful entries to ask if the participant's responses can be shared with other participants. Shared posts will be anonymous; only the age of the individual will be given.

Month one and two visits:

Participants from both groups will be asked to come to Hershey Medical Center to have their height, weight and blood pressure measured.

Month three visit:

Participants from both groups will be asked to come to Hershey Medical Center to have their height, weight and blood pressure measured. Prior to their visit, participants will be asked to complete a series of surveys online (Three-Factor Eating Questionnaire, Motivation, Weight Loss Habits, Medication log, International Physical Activity Questionnaire, Satisfaction). Participants in the control group will be given a booklet containing the writing prompts, tracking and website address to complete on their own if they so choose.

Participants will be asked if they would like to come back for an optional video interview. The interview will consist of six questions about their experience with the study.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Body mass index between 27 and 45
* E-mail and Internet access
* Able to read, write, and understand English

Exclusion Criteria:

* Weight loss of more than 5% of current body weight in previous 6 months
* Participated in weight loss research in previous 6 months
* Current use of weight loss medication or program
* History of or scheduled weight loss surgery
* Heart, liver, or kidney failure
* Been told by doctor of heart trouble
* Frequent pains in heart and chest
* Often feel faint or have spells of severe dizziness
* Bone or joint problem that has been or might be aggravated by exercise
* Physical reason for not following activity program
* History of sever cognitive impairment or major psychiatric illness
* Pregnant in previous 6 months, currently or planning to become pregnant in next 3 months
* Moving in next 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Weight | 3 months
  Weight will be measured by study staff using a Tanita BWB 800S Digital Scale.

SECONDARY OUTCOMES:
Blood Pressure | 3 months
  Blood pressure will be measured by study staff using an automatic blood pressure monitor.
Height | 3 months
  Height will be measured using a portable stadiometer.

OTHER OUTCOMES:
Sociodemographics and tobacco use | 3 months
  Age, gender, race, ethnicity, education, smoking status and other demographics will be measured by self-report
Three-factor Eating Questionnaire | 3 months
  Questionnaire asks participants about how their dietary restraint in specific circumstances
Motivation | 3 months
  Questionnaire asks participants to gauge their motivation to lose weight.
Weight Loss Habits | 3 months
  Questionnaire asks participants how often they use specific habits to lose weight
Blood Pressure Medication | 3 months
  Blood pressure medication names, doses and frequency measured by self-report
International Physical Activity Questionnaire | 3 months
  Questionnaire asks participants to estimate the frequency and duration of specific physical activities
Satisfaction Survey | 3 months
  Questionnaire asks participants about their satisfaction with specific aspects of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States